CLINICAL TRIAL: NCT06844305
Title: A Personalized, Patient-Centered Prosthetic Foot Prescription and Rehabilitation Strategy to Maximize Mobility and Satisfaction in Veterans With Lower Limb Loss
Brief Title: Personalized Prosthetic Foot Prescription and Rehabilitation for Veterans With Lower Limb Loss
Acronym: OPORP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Matthew Major, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP230014; HT9425-24-1-0319 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2025-02-15; First posted 2025-02-25 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-02

CONDITIONS: Amputation of Lower Limb
Keywords: amputation; prosthesis; prescription; physical therapy; personalized
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prosthesis Condition (Other): Participants experience walking with three prosthesis condition and select their most and least preferred.
  Interventions: Other: Prosthetic foot
- Physical Therapy (Active Comparator): Participants receive either the standard-of-care intervention (control) or an eight-week personalized physical therapy intervention.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Prosthetic foot — The most- and least-preferred prosthetic foot
  Arms: Prosthesis Condition
Other: Physical therapy — Personalized physical therapy
  Arms: Physical Therapy

SUMMARY:
The goal of clinical trial is to assess an integrated, patient-centered strategy combining user preference-based prosthetic foot prescription and subsequent targeted physical therapy to maximize satisfaction and mobility outcomes for Veterans and others with lower limb loss. The main aims it will address are:

* Assess the effect of prosthetic foot selection based on experiential preference as determined using a variable stiffness foot on mobility and satisfaction
* Assess the effect of a targeted physical therapy intervention following preference-based foot selection on mobility, balance, and satisfaction? Participants will walk with an emulator prosthetic foot to experience three different conditions that emulate different commercial feet to determine their most- and least-preferred foot. Participants' satisfaction, perceived mobility, and functional mobility will be measured and compared between their most- and least-preferred feet using the corresponding commercial feet. Participants will then be randomly assigned to receive either the standard-of-care (control group) or personalized physical therapy intervention for eight weeks using that preferred prosthetic foot. Participants' satisfaction, mobility, and balance will be measured pre- and post-intervention.

DETAILED DESCRIPTION:
Aim 1: Assess the effect of prosthetic foot selection based on experiential preference as determined using a variable stiffness foot on mobility and satisfaction. Baseline mobility and satisfaction of 50 Veterans with unilateral transtibial amputation (UTTA) will initially be evaluated with their currently prescribed prosthesis. Participants will then walk with the Variable-Stiffness Prosthetic Ankle (VSPA) Foot across real-world mobility scenarios inside and outside the laboratory. During this protocol, participants will experience three different VSPA Foot conditions that emulate different commercial feet to determine each participant's most- and least-preferred foot (with further opportunity for fine-tuning to determine the optimal stiffness category of their most preferred foot). Participants' satisfaction, perceived mobility, and functional mobility will be measured and compared between their most- and least-preferred feet using the corresponding commercial feet. Aim 2: Assess the effect of a targeted physical therapy (PT) intervention following preference-based foot selection on mobility, balance, and satisfaction. After a two-week, community-based accommodation period with their most preferred commercial foot, participants' satisfaction, perceived and functional mobility, and balance will be measured. Participants will then be randomly assigned to receive either the standard-of-care (control group) or personalized PT intervention that targets and addresses impairments in mobility and balance and patient-specific functional goals (intervention group). Following eight weeks of either standard-of-care or PT intervention, participants' satisfaction, mobility, and balance will again be measured and compared between groups (intervention vs. control) and across time periods (pre- vs. post-accommodation measurements).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation;
* At least 6 months post-amputation;
* A comfortable-fitting prosthetic socket that can be used with endoskeletal components;
* Sufficient walking abilities to safely complete study activities.

Exclusion Criteria:

* Major contralateral limb amputation LLL on the contralateral limb;
* Currently receiving physical therapy related to gait training or prosthesis use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Trinity Amputation and Prosthesis Experience Scales - Satisfaction | From enrollment (baseline) to the end of the eght week physical therapy intervention or at the time of withdrawal, whichever comes first, assessed up to 5 months
  Patient-reported outcome measure that assesses functional satisfaction with the prosthesis. The maximum value is 15 and the minimum value is 5, with higher better scores meaning a better outcome. This sum score (max 15) is used for reporting and analysis.
Prosthetic Limb Users' Survey of Mobility | From enrollment (baseline) to the end of the eght week physical therapy intervention or at the time of withdrawal, whichever comes first, assessed up to 5 months
  Patient-reported outcome measure that measures perceived mobility with a prosthesis. The maximum value is 60 and the minimum value is 12, with higher better scores meaning a better outcome. Scores are converted to t-scores for reporting and analysis.
Activities-specific Balance Confidence Scale | From enrollment (baseline) to the end of the eght week physical therapy intervention or at the time of withdrawal, whichever comes first, assessed up to 5 months
  Patient-reported outcome measure that measures perceived balance confidence. The maximum value is 60 and the minimum value is 0, with higher better scores meaning a better outcome. Scores are converted to an average through dividing the sum by number of tasks (15) for reporting and analysis.
Timed up and go | From enrollment (baseline) to the end of the eght week physical therapy intervention or at the time of withdrawal, whichever comes first, assessed up to 5 months
  Performance-based outcome measure that measures walking ability and dynamics balance. The time taken to complete the task is recorded as the score and less time means a better outcome.
Four square step test | From enrollment (baseline) to the end of the eght week physical therapy intervention or at the time of withdrawal, whichever comes first, assessed up to 5 months
  Performance-based outcome measure that measures dynamics balance. The time taken to complete the task is recorded as the score and less time means a better outcome.
Amputee Mobility Predictor | From enrollment (baseline) to the end of the eght week physical therapy intervention or at the time of withdrawal, whichever comes first, assessed up to 5 months
  Performance-based outcome measure that measures gait and balance. Each task is scored on an ordinal scale, and the maximum value is 47 and the minimum value is 0, with higher better scores meaning a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Prosthetics-Orthotics Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No